CLINICAL TRIAL: NCT02763696
Title: Establishment of a Sensitive System for Analysis of Child-bearing Women Vaginal Microbiota Which Overall Evaluation of Microscopic Precision Reference Standards
Brief Title: Establishment of a Sensitive System for Analysis of Child-bearing Women Vaginal Microbiota
Acronym: ESSACWVM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF-CRF-2015-009
Record Dates: First submitted 2016-04-26; First posted 2016-05-05 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Vaginitis
Keywords: Metagenomics; Vaginal microflora; High-throughput sequencing
MeSH Terms: conditions — Vaginitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples With DNA — Vaginal secretions from Child-bearing Women
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- normal women: Composition of Viginal flora of Child-Bearing women in normal woman
  Interventions: Other: Composition of Viginal flora of Child-Bearing women
- vaginitis women: Women of childbearing age with vaginitis
  Interventions: Other: Composition of Viginal flora of Child-Bearing women

INTERVENTIONS:
Other: Composition of Viginal flora of Child-Bearing women — Use high-throughput sequencing technology to exam Composition of Viginal flora of Child-Bearing women in different menstrual cycle and type of Vaginitis

SUMMARY:
The vaginal microbiota is an important biological barrier for host against pathogens or opportunistic pathogens. Undermining the balance of the vagina is closely related to infectious diseases and tumors.

The vaginal microbiota of child-bearing women of age is dominated by Lactobacillus species, including major four species: Lactobacillus crispatus, Lactobacillus jensenii, Lactobacillus gasseri and Lactobacillus iners, followed by obligate anaerobes such as Gardnerella vaginalis, Atopobium vaginae, Mobiluncus curtisii, and Prevotella .

Currently, There are almost 99% bacteria can not to be found with bacterial culture. Based on microscopy and conventional culture method to obtain vaginal microflora information have a variety of deviation. For this reason, The in-depth study of complex vaginal flora and the correct understanding of disease faces a serious obstacle. With the development of High-throughput sequencing technology， metagenomics can get all the composition and distribution of microorganisms from the sample which traditional knowledge may not be with microorganism culture method. Therefore, Re-evaluation of existing microflora diagnostic criteria for clinical diagnosis of the disease is necessary.

In this study, the investigators use high-throughput sequencing technology to detect women of childbearing age vaginal microflora of metagenomic distribution. Including bacteria, fungi, viruses, protozoa, and other microorganisms. Based on the study results of metagenomic, the investigators want to re-cognition the"normal flora"of women of childbearing age ,and develop vaginal microflora microscopic evaluation of the integrity of the reference standard.

ELIGIBILITY:
Inclusion Criteria:

* Normal Child-bearing Women

Exclusion Criteria:

* Pregnancy women
* Lactating women
* Using antibiotics or vaginal topical application of antibiotics over a month
* Have sexual activity in 3 days

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Child-bearing Woman
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-05-10 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The use of High-throughput sequencing to establishment a sensitive system of the composition of vaginal Microbiota of normal Child-bearing Women | From the date of first normal woman who entered the subject to a whole menstrual cycles ended up to one month
The use of High-throughput sequencing to comparison the composition of vaginal flora of normal women of childbearing age and women with vaginitis | From the date of one subjects entered to a whole menstrual cycles ended up to one month

CONTACTS AND LOCATIONS:
Overall Officials: Yawen Wang, Ph.D, Study Chair — First Affiliated Hospital of Xian Jiaotong University
Locations (1):
- First Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided